CLINICAL TRIAL: NCT05112302
Title: Use of Virtual Reality as an Adjunct for Anesthesia During Orthopedic Procedures Under Regional or Central Neuraxial Nerve Block. A Pilot and Feasibility Study
Brief Title: A Study to Evaluate Virtual Reality As Adjunct to Anesthesia During Orthopedic Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Klaus D. Torp, Principal Investigator, Mayo Clinic
Other Study IDs: 21-005305
Record Dates: First submitted 2021-10-13; First posted 2021-11-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Knee Arthropathy; Hip Injuries
Keywords: virtual reality; knee arthroplasty; hip arthroplasty
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Virtual reality
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: Virtual reality — Use of virtual reality goggles during procedure

SUMMARY:
The purpose of this study is to obtain feedback from patients and orthopedic surgeons who agree to use virtual reality (VR ) as an adjunct to standard of care in orthopedic cases under regional or central neuraxial nerve block. This will serve as a preliminary study for future trials to compare outcomes between VR and standard of care vs standard of care only.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Patients scheduled for orthopedic procedure under regional or central neuraxial nerve block (anterior primary hip arthroplasty or primary knee arthroplasty).
* Subject willing to participate and able to provide informed consent.

Exclusion Criteria:

* Age < 18 years old.
* History of motion sickness or blindness.
* Unable to consent due to cognitive difficulty.
* Current diagnosis of epilepsy, dementia, or other neurological disease that may prevent use of VR hardware and software.

Sensitivity to flashing light or motion.

* Recent stroke.
* Injury to the eyes, face, neck, or arms that prevents comfortable use of VR hardware or software, or safe use of the hardware (e.g., open wound, sores, or skin rash on face).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective orthopedic surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Impact of virtual reality on anxiety level | Up to 2 hours
  Evaluate patients' satisfaction with using virutal reality and reduction in anxiety during orthopedic procedures

SECONDARY OUTCOMES:
Impact of virtual reality on pharmacological therapy doses | Up to 2 hours
  Elucidate the impact of VR on pharmacological therapy doses required for proper analgesia and anxiolysis and on reduction of drug side effects in patient using VR during surgeries.
Impact of virtual reality on patient's perioperative temperature | Up to 3 hours
  Evaluate if utilizing virtual reality has a positive impact in preventing patient hypothermia intra- and post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Torp, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jackson, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials